CLINICAL TRIAL: NCT04446065
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Clinical Trial to Protect Health Workers Against COVID-19 by Using Previfenon® as Chemoprophylaxis During a SARS-CoV-2 Outbreak. The HERD Study
Brief Title: Previfenon® as Chemoprophylaxis of COVID-19 in Health Workers
Acronym: HERD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MELISA Institute Genomics & Proteomics Research SpA (Industry)
Collaborators: Universidad Austral (Unknown)
Responsible Party: Principal Investigator, Elard Koch, PhD, Head of Reserach, MELISA Institute Genomics & Proteomics Research SpA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEL109042020
Record Dates: First submitted 2020-06-23; First posted 2020-06-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; SARS-CoV2
Keywords: clinical trial; chemoprophylaxis; coronavirus; antiviral agents; epigallocatechin-3-gallate
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — epigallocatechin gallate; Starch

STUDY DESIGN:
Intervention Model Description: The study will use 2 parallel groups in each center to compare the effects of an oral formulation of EGCG (Previfenon®, patent pending) with those of placebo (starch) in the prevention of respiratory disease caused by SARS-CoV-2 (COVID-19) in health care workers directly exposed to clinical care, daily contact, or traffic of individuals with suspected for COVID-19 during the epidemic outbreak.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Previfenon® (Experimental): Participants will receive coded non-transparent bottles of Previfenon®, each containing 90 EGCG capsules (250 mg per capsule plus excipients) The total EGCG dose per patient will be 750 mg/day (3 capsules) for 40 consecutive days as minimum or a maximum variable time between 60 to 70 days. It will be divided into three daily intakes of one capsule of Previfenon® every 8 hours.
  Interventions: Drug: Previfenon®
- Placebo (Placebo Comparator): Participants will receive coded non-transparent bottles of placebo, each containing 90 starch capsules (250 mg plus excipients) under the same dosage, frequency and duration that Previfenon@ arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Previfenon® — Every capsule of Previfenon® (patent pending) provides 250 mg EGCG ≥ 98% purity with a carefully selected set of excipients to improve flowability, stabilize EGCG against early auto-oxidation, and increase its hepatoprotective activity with prolonged use.
  Other Names: Epigallocatechin-3-Gallate, EGCG
  Arms: Previfenon®
Drug: Placebo — Participants will receive placebo starch capsules (250 mg plus excipients) identical in appearance and taste to Previfenon® capsules in a double-blind manner.
  Other Names: Starch
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to determine the efficacy of Previfenon® (EGCG) to prevent COVID-19, enhance systemic immunity, and decrease the frequency and intensity of selected symptoms when used as pre-exposure chemoprophylaxis to SARS-CoV-2.

DETAILED DESCRIPTION:
Background. Experimental studies have revealed that epigallocatechin-3-galeate (EGCG), a biologically active polyphenol extracted and purified from Camellia Sinensis, may prevent infection by various kinds of viruses, including coronaviruses. Recent double blind, placebo controlled clinical trials, reported up to 75% reduction in the risk of respiratory infection by healthcare workers during an outbreak of H1N1 influenza, simultaneously enhancing systemic immunity by increasing proliferation of ϒδ T cells (28%) and production of IFN-γ (26%). In molecular docking studies against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2, the causal agent of coronavirus disease 2019 outbreak also known as COVID-19) EGCG was identified as a candidate with very high potential for antiviral chemoprophylaxis of COVID-19.

Primary objective: To determine whether Previfenon®, a proprietary formulation of EGCG ≥ 98% purity stabilized with selected excipients, may clinically prevent COVID-19, enhance systemic immunity, decrease the rate for acute respiratory disease, and reduce the frequency and intensity of selected symptoms of COVID-19.

Secondary objective: To determine safety and tolerability of Previfenon® in terms of liver toxicity and frequency of adverse events.

Design. Multicenter randomized double-blind placebo-controlled trial of healthcare workers in treatment by 40 consecutive days as minimum, or a maximum variable time between 60 to 70 days during a SARS-CoV-2 outbreak in Latin American hospitals exposed to clinical care, contact, or circulation of patients with suspected respiratory acute disease caused by SARS-CoV-2 also known as COVID -19.

Sample size: A minimum effect size of 25% (OR = 0.75) is considered; 5% alpha error; 90% power; R = 0.25 for confounders and 20% for loss to follow up. If a conservative event rate of 7.5% in the untreated group is considered, the trial will require 524 participants (262 each group); if the event rate reaches 13.5%, the trial will require 298 participants (149 each group). It is expected to recruit between 100 to 240 subjects per site.

Intervention. The treatment group will receive 3 capsules of Previfenon® daily containing 250 mg of EGCG one every 8 hours. The control group will receive 3 placebo capsules (starch 250 mg) under the same frequency.

Outcomes. The primary outcome will be the rate of clinically defined COVID-19 confirmed with rt-PCR for SARS-CoV-2 viral RNA. Secondary outcomes will be (1) rate of positive cases for IgM or IgG anti-SARS-CoV-2 as measured by a rapid immuno-chromatographic test; (2) rate of positive cases for rtPCR for SARS-Cov-2 viral RNA (3) rate of hospitalization for acute respiratory disease; (4) total rate of lower or upper acute respiratory disease. Exploratory outcomes will be the frequency and intensity of selected symptoms for COVID-19. Safety outcomes will be the number of events of major hepatic toxicity accounted by an increment in liver enzymes and frequency of adverse events during the treatment.

Analysis. Comparison of frequencies, means, and proportions for all relevant variables between treated group and placebo will be performed. An interim analysis will be conducted with the first 366 subjects with at least 20 days of treatment during the outbreak. It will be utilized logistic regression to explore the ongoing effect size in a fixed-effect model. Disease-free person-days curves over the total follow up period will be analyzed using Kaplan-Meier and the total effect size will be computed by Cox proportional hazards multiple regression.

Leading hypothesis: The use of Previfenon® will have a high efficacy in the chemoprophylaxis of COVID-19 through multiple complementary mechanisms, which ultimately prevent an efficient incubation of the SARS-CoV-2 in the host cells, and simultaneously, enhances systemic immunity against the pathogen.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer healthcare worker with any valid credential of the center
* 25 years old and over
* Not having been diagnosed with COVID-19
* A healthy individual as per investigator's judgment or stating stable non-transmissible chronic disease without hospitalization in the last year, without change of medications or addition of medications to treat chronic illnesses in the last 3 months.
* No pregnancy or breastfeeding
* Female subjects of childbearing potential using an effective family planning method or surgical sterilization or not sexually active during the study
* Do not drink more than 300 ml of tea a day
* Do not take supplements or products containing EGCG during the study
* Being able to set aside time each day to complete the study questionnaires
* Being able to read and understand the informed consent form before the study

Exclusion Criteria:

* Healthcare worker who does not have a valid credential from the center
* Under 25 years of age
* Having been diagnosed with a positive rtPCR for COVID-19
* History of febrile acute respiratory disease within the previous 12 weeks
* Volunteer with significant alteration from laboratory tests (standard biochemical profile and hemogram) at screening. A significant abnormality will be defined according investigator's medical judgment.
* Women during pregnancy or breastfeeding
* Female subjects of childbearing age who are sexually active during the study who do not use an effective method of family planning or do not have surgical sterilization
* Known allergy to green tea or EGCG
* Known starch allergy
* User of any medication or supplement containing EGCG
* Volunteer using immunosuppressive drugs
* Autoimmune disease (Lupus, Sjögren or another), liver disease
* Anemia requiring treatment
* Having a chronic infectious disease under treatment

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Event of clinical acute respiratory disease with a diagnosis of COVID-19 confirmed with rtPCR | The date for censoring a case will be defined as that date when the rtPCR test results positive minus 4 days, with the aim to calculate the time free of clinically defined COVID-19 infection over 40 to 70 days of intervention
  A positive case or event of COVID-19 is defined as a patient with acute respiratory illness presenting fever (37.8º C); at least one of the following symptoms: odynophagia, cough, myalgia, or dyspnea; and a specific positive rtPCR test for SARS-CoV-2.

SECONDARY OUTCOMES:
Rate of positive cases for IgM and IgG anti-SARS-CoV-2 | Positive cases in each two-week examination and to the end of the study over 40 to 70 days of intervention
  Rate of positive cases for IgM and IgG anti-SARS-CoV-2 measured by immunochromatographic test in treatment and placebo group at the end of the study
Composite outcome considering symptomatic and asymptomatic cases with positive rtPCR test | Positive cases in each two-weeks examination and to the end of the study over 40 to 70 days of intervention
  Rate of asymptomatic cases defined as a positive rtPCR for SARS-CoV-2 viral RNA but with no symptoms of COVID-19 in treatment and placebo group at the end of the study, and a composite outcome considering symptomatic and asymptomatic cases (i.e. all cases with positive rtPCR test)
Hospitalization due to any acute respiratory infection | Positive cases in each two-week examination visit and to the end of the study over 40 to 70 days of intervention
  Rate of hospitalizations due to any acute respiratory infection at the end of the study
Event of upper and lower airway respiratory infection | Positive cases in each two-week examination and to the end of the study over 40 to 70 days of intervention
  Global frequency of events of upper and lower airway respiratory infections

OTHER OUTCOMES:
Exploratory outcome: Frequency and intensity of selected symptoms for COVID-19 | Different VAS scores calculated each two-week examination visit over 40 to 70 days of intervention
  Registry of Visual Analogue Scale (VAS) in the log diary of every healthcare worker for the following selected symptoms: cough, muscle pain (myalgia); difficulty breathing (dyspnea); loss of smell (anosmia); loss of taste (ageusia); pain when swallowing (odynophagia, sore throat); and finally headache
Primary safety outcome: event of major hepatic harm | Cases accounted by liver profile lab test in each two-week examination visit over 40 to 70 days of intervention.
  Elevation of liver enzymes over 5 times the normal value
Event of liver enzymes over 3 times the normal value | Cases accounted by liver profile lab test in each two-week examination visit over 40 to 70 days of intervention
  Elevation of liver enzymes over 5 times the normal value
Frequency of adverse events | Records of self-reported adverse effects on log dairy accounted in each examination visit over 40 to 70 days of intervention
  Any adverse event reported over the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Elard S Koch, PhD, Study Director — MELISA Institute Genomics & Proteomics Research SpA

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be published as open access article and all IPD that underlie results in a publication will be shared, preferentially as supplementary data set or available in a public repository. Any sensitive personal data/information will be not included.
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: MELISA Institute — http://www.melisainstitute.org